CLINICAL TRIAL: NCT06329128
Title: Evaluation of the Effectiveness of Manual Therapy in Patients With Knee Osteoarthritis: Randomized Controlled Single-blind Clinical Study
Brief Title: Evaluation of the Effectiveness of Manual Therapy in Patients With Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba GÖNEN, Assistant Professor, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/04
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Manual therapy; Exercise; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Participants were divided in two groups. One groups will get electrotherapy, exercise(home programme) and manuel therapy intervention. One group will be the control group. Control group will get electrotherapy and exercise (home programme).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): This group will get manuel therapy that combinated electroterapy and hm programme (exercise).
  Interventions: Other: Experimental: Study Group
- Control Group (Active Comparator): This group will get traditional therapy (electrotherapy and exercise)
  Interventions: Other: Active Comparator: Control Group

INTERVENTIONS:
Other: Experimental: Study Group — A 15-session (5 days a week / 3 weeks) physiotherapy and rehabilitation (electrotherapy and home program) program will be applied to both groups.
  Electrotherapy application; It will consist of Hotpack (15 minutes), TENS (20 minutes), Ultrasound (10 minutes) applications. For the home program, a program consisting of isometric and isotonic exercises will be given to the muscles around the knee. The home program will be followed with an exercise diary.
  In the manual therapy group, in addition to the above treatment, manual therapy will be given 3 days a week. The content of the manual therapy program is as follows;
  * Patellofemoral joint superior-inferior mobilization
  * Medial-lateral mobilization with active knee flexion
  * Tibiofemoral joint ventral (anterior-posterior) mobilization
  * Tibiofemoral traction mobilization
  Arms: Study Group
Other: Active Comparator: Control Group — A 15-session (5 days a week / 3 weeks) physiotherapy and rehabilitation (electrotherapy and home program) program will be applied to both groups.
  Electrotherapy application; It will consist of Hotpack (15 minutes), TENS (20 minutes), Ultrasound (10 minutes) applications. For the home program, a program consisting of isometric and isotonic exercises will be given to the muscles around the knee. The home program will be followed with an exercise diary.
  Arms: Control Group

SUMMARY:
The aim of this study is to investigate the effects of three different applications (Manual therapy, electrotherapy and home program) on long-term pain, joint range of motion and, secondarily, the functional level of the knee.

DETAILED DESCRIPTION:
Osteoarthritis (OA); It is a chronic degenerative joint disorder characterized by joint pain, stiffness, decreased range of motion and muscle weakness. The main goal of healthcare professionals is to control the pain that increases with the gradually decreasing quality of life and to improve functions as a result. Conservative treatments include medical approaches as well as methods with demonstrated therapeutic effects such as exercise and physical activity. Exercise plays an important role in the management of chronic disabling disease. Looking at systematic reviews, there is high evidence that exercise reduces pain and improves physical function in patients with knee osteoarthritis. Manual therapy approaches have also been used recently to inhibit movement limitation and pain in the joint, and studies showing their benefits are increasing. The American College of Rheumatology has stated that it is beneficial to add manual therapy sessions to individual exercises in rehabilitation methods for patients. In terms of physiotherapy approaches in OA, electrotherapy modalities with low evidence are used. Among these modalities, the effects of TENS and Ultrasound are the most studied applications. Although the effects of TENS compared to placebo have been shown, there are also opposite results regarding TENS and ultrasound applications. There are many studies in the literature comparing types of manual therapy and investigating their combination with exercise. Some studies have demonstrated the effects of combining exercise treatments with a manual therapy program in improving pain and function. A recent study showed that patients who participated in an MT program had improved functional level compared to those who did not receive MT, but exercise therapy alone was superior in improving performance-based functional scores. A few studies comparing manual therapy with electrotherapy have been conducted recently. In this study, TENS and cold application were shown to be ineffective in improving pain, joint stiffness and physical functions compared to manual therapy in patients with OA. While manual therapy can reduce pain in OA thanks to its neurophysiological effects, it also aims to correct the changed arthrokinematics by restoring the optimal kinematics between joint accessory mobility and joint surfaces. Taylor et al. showed that the combination of exercise and extension mobilization applied in a single session can reduce end-range rotational stiffness. However, in the applications, comparisons are made between manual therapy and exercise combination or manual therapy and electrotherapy modalities. To our knowledge, there is no study in the literature comparing three different applications. Therefore, we hypothesized that manual therapy would be more effective than electrotherapy modalities and a home program in the long term in patients with knee OA. The aim of this study is to investigate the effects of three different applications (Manual therapy, electrotherapy and home program) on long-term pain, joint range of motion and, secondarily, the functional level of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee osteoarthritis according to the clinical and radiological diagnostic criteria of the American College of Rheumatology
* Patients with osteoarthritis stage II or III according to the Kellgren-Lawrence classification

Exclusion Criteria:

* Having had knee surgery or lower extremity surgery
* Those who have received any physical therapy program in the last week
* Those with serious arrhythmia or a pacemaker
* Inflammatory arthritis or neuromuscular
* Having a history of malignancy
* Pregnant
* Those with open wounds and infections in the knee area
* Those with severe hypoesthesia or neurological disease
* Those with bleeding conditions and thrombophlebitis

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female individuals who agree to participate in the study will be included.
Enrollment: 40 (Estimated)
Dates: Start 2024-03-25 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The pain | through of the study, average 5 weeks and 3 months later
  Mc Gill Short Form will used to determine the type and severity of the pain. A short form of the McGill Pain Questionnaire (SF-MPQ) has been developed. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Functional status | through of the study, average 5 weeks and 3 months later
  Western Ontario ve McMaster Universities (WOMAC) index will used to determine the knee osteoarthritis functional status. The questionnaire, developed at Western Ontario and McMaster University in 1982, includes a total of 24 items consisting of the subparameters Pain (5), Stiffness (2), and Physical function (17). Scoring of the items is done according to the Likert scale. The degree of pain and strain is indicated by giving points from 0 to 4 on the Likert scale. The total score is calculated as a percentage by multiplying the score by 100 and dividing by 96, which is the maximum total score.
The quality of Life | through of the study, average 5 weeks and 3 months later
  Nothingham Health Profile will used to determine the quality of life. Hunt et al. NHP, which was developed in 1981 and used to evaluate the quality of life, consists of 2 subsections. Part 1 includes the subparameters of Pain, Emotional Reactions, Sleep, Social Isolation, Physical Activity and Energy, and Part 2 measures the frequency of health-related problems in work and home life, hobbies, social and sexual life. Part 1 is measured between 0-600 points, and Part 2 is measured between 0-7 points. As the score increases, the quality of life decreases
Lower extremity functional strength and balance test | through of the study, average 5 weeks and 3 months later
  Sit to stand test will used to determine Lower extremity strength and balance. The sit to stand test, which evaluates lower extremity muscle strength and endurance and is frequently used in osteoarthritis patients, is performed on a chair without armrests with a height of approximately 44 cm. The patient sits in the middle of the chair with his back straight. Feet touch the ground approximately shoulder-width apart, with one foot slightly in front of the other to help maintain balance. Arms are crossed on the shoulders and the patient is asked to stand up and sit like this for 30 seconds. Sitting and standing for less than 10 repetitions after 30 seconds indicates lower extremity weakness.
Functional mobility | through of the study, average 5 weeks and 3 months later
  Time up and go test will used to determine functional mobility. Time up and go test was developed by Podsiadlo et al. in 1991. It was developed by Mathias et al. as a modification of the Get-Up and Go Test. For performance measurement that evaluates fall risk and functional mobility, a 3-meter area is determined in front of the chair. The patient is asked to get up from the chair, walk a distance of 3 meters, and then come back and sit on the chair. Time is measured in seconds with a stopwatch. It is determined that there is a risk of falling when the test is completed in more than 12 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson AE, Allen KD, Golightly YM, Goode AP, Jordan JM. A systematic review of recommendations and guidelines for the management of osteoarthritis: The chronic osteoarthritis management initiative of the U.S. bone and joint initiative. Semin Arthritis Rheum. 2014 Jun;43(6):701-12. doi: 10.1016/j.semarthrit.2013.11.012. Epub 2013 Dec 4. PMID 24387819
- [Background] Zeng C, Li H, Yang T, Deng ZH, Yang Y, Zhang Y, Ding X, Lei GH. Effectiveness of continuous and pulsed ultrasound for the management of knee osteoarthritis: a systematic review and network meta-analysis. Osteoarthritis Cartilage. 2014 Aug;22(8):1090-9. doi: 10.1016/j.joca.2014.06.028. Epub 2014 Jul 4. PMID 24999112
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Rutjes AW, Nuesch E, Sterchi R, Kalichman L, Hendriks E, Osiri M, Brosseau L, Reichenbach S, Juni P. Transcutaneous electrostimulation for osteoarthritis of the knee. Cochrane Database Syst Rev. 2009 Oct 7;2009(4):CD002823. doi: 10.1002/14651858.CD002823.pub2. PMID 19821296
- [Background] Conaghan PG, Kloppenburg M, Schett G, Bijlsma JW; EULAR osteoarthritis ad hoc committee. Osteoarthritis research priorities: a report from a EULAR ad hoc expert committee. Ann Rheum Dis. 2014 Aug;73(8):1442-5. doi: 10.1136/annrheumdis-2013-204660. Epub 2014 Mar 13. PMID 24625626
- [Background] Zasadzka E, Borowicz AM, Roszak M, Pawlaczyk M. Assessment of the risk of falling with the use of timed up and go test in the elderly with lower extremity osteoarthritis. Clin Interv Aging. 2015 Aug 7;10:1289-98. doi: 10.2147/CIA.S86001. eCollection 2015. PMID 26300633
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] Courtney CA, Witte PO, Chmell SJ, Hornby TG. Heightened flexor withdrawal response in individuals with knee osteoarthritis is modulated by joint compression and joint mobilization. J Pain. 2010 Feb;11(2):179-85. doi: 10.1016/j.jpain.2009.07.005. Epub 2009 Nov 27. PMID 19945353